CLINICAL TRIAL: NCT02028611
Title: Comparison of Gray-scale Inverted Rib Series With Conventional Ones in Rib Fracture Detection by Emergency Physicians and Medical Students
Status: Completed | Type: Observational
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Joonbum Park, MD, Hanyang University
Other Study IDs: JPark
Record Dates: First submitted 2013-08-28; First posted 2014-01-07 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Rib Fracture
Keywords: Rib fracture; Inverted grayscale
MeSH Terms: conditions — Rib Fractures

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional

SUMMARY:
There were many studies which examined the availability of inverted gray-scale chest X-ray for increasing the detection of lung nodules. In emergency medicine, rib fracture is an important part for patient's disposition, so investigators designed this study to evaluate the availability of inverted gray-scale chest X-ray for the detection of rib fracture.

ELIGIBILITY:
Inclusion Criteria:

* Emergency resident who want to participate

Exclusion Criteria:

* Emergency resident who does not want to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Emergency medicine residents
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Sensitivity of detection for rib fracture | up to 12 weeks
  Sensitivity of detection for rib fracture in 139 fracture of 55 patients

SECONDARY OUTCOMES:
Accuracy for rib fracture | up to 12 weeks

REFERENCES:
- [Derived] Park JB, Cho YS, Choi HJ. Diagnostic accuracy of the inverted grayscale rib series for detection of rib fracture in minor chest trauma. Am J Emerg Med. 2015 Apr;33(4):548-52. doi: 10.1016/j.ajem.2015.01.015. Epub 2015 Jan 20. PMID 25690384